CLINICAL TRIAL: NCT05998538
Title: Patients With Higher BMI Produces More Postoperative Drainage Volume and Longer Length of Stay in Cross-Sectional Study: a Comparison of Total vs Partial Knee Arthroplasty
Brief Title: Patients With Higher BMI Produces More Postoperative Drainage Volume and Length of Stay in Cross-Sectional Study
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ludwig Andre Pontoh, DR, Indonesia University
Other Study IDs: 23082020
Record Dates: First submitted 2023-08-09; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TKA (Total Knee Arthroplasty) procedure: Total Knee Arthroplasty
  Interventions: Procedure: Knee Replacement
- UKA (Uni Knee Arthroplasty) procedure: Uni Knee Arthroplasty
  Interventions: Procedure: Knee Replacement

INTERVENTIONS:
Procedure: Knee Replacement — Total vs Partial Knee Replacement

SUMMARY:
Partial knee arthroplasty theoretically produces less blood loss compared to total knee arthroplasty (TKA) due to a lesser invasive procedure. Medial unicompartmental knee arthroplasty (UKA) is the most common partial knee arthroplasty performed due used due to the most commonly impacted medial knee. This study compared the postoperative drainage volume and length of stay (LOS) of TKA vs UKA and evaluated its comparison with patient characteristics.

DETAILED DESCRIPTION:
Theoretically, UKA will produce less blood loss due to a shorter skin incision, quadriceps sparing muscle approach, persistence of cruciate ligaments, and less femorotibial dislocation.7 However, studies investigating drainage volume in UKA are still limited. In this study, we compared the drainage volume of patients undergoing TKA vs UKA and evaluated several parameters that contributed the production. This study has not received any funding or grant.

ELIGIBILITY:
Inclusion Criteria:

* grade 4 Osteoarthritis

Exclusion Criteria:

* previous trauma
* infection
* blood coagulation disorder

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: medical records of patients who underwent primary TKA and UKA between December 2019 and October 2022
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Drainage Volume | 3-5 days post op
  total drainage volume

SECONDARY OUTCOMES:
LOS | pre-op until drainage removed, 3-6 days post op
  length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Ismail H Dilogo, Prof, Study Director — Indonesia University
Locations (1):
- Pondok Indah Hospital, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No